CLINICAL TRIAL: NCT00189046
Title: Effects of Pain on Driving Performance, Attentional Capacity and Psychomotor Performances: a Comparative Study Between Healthy Controls and Chronic Pain Patients.
Brief Title: Effects of Pain on Driving Performance and Cognition.
Status: Terminated | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: Utrecht University (Other)
Other Study IDs: 03/237-E
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2004-12

CONDITIONS: Chronic Pain
Keywords: driving, chronic pain, attention
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

INTERVENTIONS:
Behavioral: driving and laboratory tests

SUMMARY:
It has been suggested that cognitive functioning is impaired in chronic pain patients. Since most of these pain patients engage in daily activities including driving, it was hypothezised that they may have an increased risk of becoming involved in traffic accidents.

DETAILED DESCRIPTION:
Most chronic pain patients engage in daily activities including driving. Driving a car is a complex task requiring mental alertness and a variety of cognitive functions such as perception, attention, learning, memory and decision making.Several studies have demonstrated cognitive impairments on laboratory tasks in patients with chronic pain, particularly on measures assessing attentional capacity, processing speed and psychomotor speed. These findings suggest that car driving performance might be impaired, and that chronic pain patients may therefore have an increased traffic accident risk. Unfortunately, no studies have investigated the impact of chronic pain on actual driving ability. The present study was designed to investigate the effects of chronic pain on actual driving performance during normal traffic. In addition to the on-the-road driving test, psychomotor, and memory tests measuring driving-related skills were conducted in the laboratory. Moreover, effects of pain on an attentional capacity test were tested using event-related potentials.

ELIGIBILITY:
Inclusion Criteria:

age driving licence driving experience normal vision right-handed fluently Dutch speaking

Exclusion Criteria:

psychological or physical disorder drug or alcohol abuse psychotropic medication use excessive smoking, drinking

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30
Dates: Start 2004-01; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Overall Officials: Edmund Volkerts, PhD, Principal Investigator — University of Utrecht, Department of Psychopharmacology
Locations (1):
- Department of Psychopharmacology, Utrecht, Utrecht, Netherlands